CLINICAL TRIAL: NCT06341218
Title: The Effect Of Simulation-Supported Pediatric Cardiopulmonary Resuscitation Training Based On Crew Resource Management On Knowledge, Attitude, And Performance
Brief Title: The Effect Of Simulation-Supported Pediatric CPR Training Based On CRM On Knowledge, Attitude, And Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zonguldak Bulent Ecevit University (Other)
Collaborators: Ege University (Other)
Responsible Party: Principal Investigator, Signem ANOL KILIÇ, research assistant, Zonguldak Bulent Ecevit University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 21-5T/3
Record Dates: First submitted 2023-11-28; First posted 2024-04-02 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-04

CONDITIONS: Cardiopulmonary Resuscitation
Keywords: crew resource management; cpr; multidisciplinary health team; pediatric nursing; patient simulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The intervention group was divided into 5 CPR teams consisting of 5 nurses and 2 physician assistants. While forming the intervention group, stratified random sampling was performed by targeting the years of professional experience of assistant physicians and nurses and homogeneity between subgroups was ensured. CRM-Based Pediatric CPR Training was given to the intervention group.
  Interventions: Other: Pediatric Cardiopulmonary Resuscitation Training Based On Team Resource Management
- Control Group (No Intervention): The Control group was divided into 5 CPR teams consisting of 5 nurses and 2 physician assistants. While forming the control group, stratified random sampling was performed by targeting the years of professional experience of assistant physicians and nurses, and homogeneity between subgroups was ensured. The control group was assumed to know pediatric CPR management as per their clinical duties and no educational intervention was made.

INTERVENTIONS:
Other: Pediatric Cardiopulmonary Resuscitation Training Based On Team Resource Management — The sociodemographic information form, Pediatric CPR knowledge level and teamwork attitudes pretest were administered to the healthcare teams just before the training intervention.
  The intervention group received a 3-hour training intervention on technical/non-technical skills for CRM-Based Pediatric CPR Training To measure pediatric CPR team performance, 5 different scenarios were prepared by the researcher by INACLS standards. One day after the training intervention, simulation application including pediatric cardiac arrest scenarios was applied to all CPR teams in the intervention(5 groups) and control(5 groups) groups. The scenario content was based on a 5-year-old male patient diagnosed with Pneumonia+Septic Shock.
  Pediatric CPR skill levels of the healthcare teams were evaluated during the simulation practice. Immediately after the simulation, the post-intervention post-test of Pediatric CPR knowledge level and team attitudes of the healthcare teams was performed.
  Arms: Intervention Group

SUMMARY:
Crew Resource Management is a training system that aims to use all available resources effectively and increase safety by improving technical knowledge and skills as well as non-technical skills in risky tasks such as CPR. In safe critical patient management, the healthcare team should have interpersonal skills such as communication, stress management, teamwork, and leadership, cognitive skills such as situational awareness, task completion, planning, monitoring the situation, and rapid response to critical incidents, in addition to technical skills. To improve outcomes after pediatric cardiac arrest, many systems have been developed for performance measurement and quality improvement initiatives of the healthcare team. However, studies are needed to evaluate the effects of these systems. This study was planned to evaluate the effectiveness of simulation-supported pediatric cardiopulmonary resuscitation training based on team resource management on knowledge, attitude, and performance of the healthcare team in the pediatric intensive care unit.

DETAILED DESCRIPTION:
The study was conducted to evaluate the effectiveness of simulation-supported pediatric cardiopulmonary resuscitation training based on the principles of Team Resource Management (ERM) on the knowledge, attitude, and performance of the healthcare team in the pediatric intensive care unit.

In this prospective randomized controlled study, nurses and physician assistants working in the Pediatric Intensive Care Unit (n=35), determined as the intervention group, and in the Pediatric Emergency Department (n=35), which was determined as the control group, were included in the sample. The intervention group received EKY-based pediatric CPR training, and it was assumed that the control group knew pediatric CPR management by their clinical duties. All CPR teams in the intervention and control groups were simulated with pediatric cardiac arrest scenarios and their pediatric CPR knowledge, attitudes, and performance were examined.While forming the intervention and control groups, stratified random sampling was performed by targeting the years of pediatric professional experience of resident physicians and nurses, and homogeneity between the groups was ensured.

The intervention group received CRM based pediatric CPR training and the control group was assumed to know pediatric CPR management as per their clinical duties. 'Healthcare Team Socio-Demographic Data Collection Form', 'Pediatric CPR Information Form', 'Teamwork Attitudes Scale', 'Pediatric CPR Team Performance Checklist', 'Student Satisfaction in Learning and Self-Confidence Scale' was used to collect the data for the study.

ELIGIBILITY:
Inclusion Criteria:

* Working in Ege University Pediatric Intensive Care Unit or Pediatric Emergency Service
* Voluntary acceptance to participate in the study
* Participated in CPR case management at least once
* Not having received ECM training before
* Not having received any training on Pediatric CPR and ECPR during the implementation phase of the study

Exclusion Criteria:

* Voluntary refusal to participate in the study,
* Never participated in CPR case management,
* Having received EKY training before,
* Having received any training in Paediatric CPR and ECM during the implementation phase of the study,
* Incomplete completion of the data collection tools of the study or failure to complete the simulation phase

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2021-02-25 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
Socio-demographic data of the healthcare team | Baseline
  In this form, there are closed-ended questions about the participant's age, gender, occupation, educational status, duration of professional experience, area of professional experience, the status of receiving Pediatric CPR training in undergraduate education, the status of attending the Pediatric CPR Course, and the status of participating in CPR case management in the clinic.
  In addition, open-ended questions were included to evaluate the reasons for the difficulties experienced in the management of the CPR process, the perception of a functional team in CPR management, the status of providing functional teamwork in risky tasks such as CPR in their clinics, and what are the individual-clinical-organizational suggestions to improve ECM management in the CPR process.
Pediatric KPR knowledge level | 2 month
  The effect of simulation-supported pediatric KPR training based on team resource management on knowledge
  The form includes a total of 25 statements, including 13 true and 12 false statements for the management of the Pediatric CPR process. A cut-off point of 80 points was set for the participants to be evaluated as successful in the form in which the level of knowledge of the participants was determined. For each statement in the form, the participants were expected to answer as 'True' - 'False' - 'No Idea'; each item was evaluated over 4 points.
Pediatric KPR team attitude level | 2 month
  The effect of simulation-supported pediatric KPR training based on team resource management on team attitude
  The Teamwork Attitudes Scale includes 5 sub-dimensions (team structure, leadership, situation monitoring, mutual support, and communication) and 28 items. The scale is a 5-point Likert-type scale (Strongly Disagree=1 point, Disagree=2 points, Undecided=3 points, Agree=4 points, Strongly Agree=5 points). As a result of the evaluation of the scale total score averages and sub-dimension score averages, the highest score is 140 and the lowest score is 28. As a result of the evaluation of the scale, the high score of the individual shows that the teamwork attitude is positive.
Pediatric KPR team performance level | 2 month
  The effect of simulation-supported pediatric KPR training based on team resource management on performance
  Pediatric CPR Team Performance Checklist; while the participant performed the skill expected from him/her in the simulation environment, the researcher monitored how this skill was performed and evaluated through pre-structured and progressive checklists. In the evaluation of the Pediatric CPR Team Performance Checklist; according to the performance of the participant, each item was evaluated as 'Not Performed=0 points', 'Partially Performed=1 point', and 'Performed=2 points'. Total score averages were used in the evaluation. The Pediatric CPR Team Performance Checklist includes the following sections; Phase 1: Pre-CPR Performance Checklist (16 items) Phase 2: CPR Process Performance Checklist (16 items) Phase 3: Post-KPR Performance Checklist (6 items) Phase 4: CPR Process Non-Technical Skills Checklist (13 items)

CONTACTS AND LOCATIONS:
Overall Officials: SİĞNEM ANOL KILIÇ, PhD, Principal Investigator — Research assistant
Locations (1):
- Ege University, Izmir, Bornova, Turkey (Türkiye)